CLINICAL TRIAL: NCT01516788
Title: Photoprovocation Testing in Subjects With Cutaneous Lupus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 814860
Record Dates: First submitted 2012-01-12; First posted 2012-01-25 (Estimated); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Lupus Erythematosus; Photosensitivity Conditions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phototesting (Experimental)
  Interventions: Other: Phototesting

INTERVENTIONS:
Other: Phototesting — Single MED dose on Day 2

SUMMARY:
Photosensitivity is well documented among lupus patients and is one of the diagnostic criteria for systemic lupus erythematosus (SLE). Photosensitivity is highly prevalent in lupus and has a wide range of clinical presentations. However, photosensitivity is a poorly defined in lupus and its pathogenesis is not well understood. The purpose of this study is to characterize the early clinical and histopathological changes in lupus skin that occur as a response to ultraviolet light.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have a diagnosis of CLE based on either the Gilliam classification of DLE and SCLE, or SLE based on the American College of Rheumatology criteria.

Exclusion Criteria:

1. Participants who do not meet criteria for either CLE or SLE.
2. Participants with a diagnosis of Erythropoietic Protoporphyria and Solar Urticaria, or another photodermatoses other than Polymorphous light eruption.
3. Participants who are not yet 18 years old or who are not capable of giving written informed consent prior to enrolling in the study.
4. Participants who have undergone any recent phototesting, or phototherapy exposure, or those who are suspected of having a drug-induced photosensitivity.
5. Female participants who are pregnant or breastfeeding will be excluded from the study. This will be determined by patient self-reporting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-12; Primary Completion 2018-07-02 (Actual); Study Completion 2018-07-02 (Actual)

PRIMARY OUTCOMES:
The change from baseline of the neutrophil and inflammasome response to ultraviolet radiation at 24 hours. | 24 hours and 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States